CLINICAL TRIAL: NCT03495297
Title: A Prospective Randomised CompArative Trial of SubcutanEous ImplanTable CardiOverter-DefibrillatoR ImplANtation With and Without DeFibrillation Testing
Brief Title: A Randomised Trial of S-ICD Implantation With and Without Defibrillation Testing
Acronym: PRAETORIAN-DFT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Principal Investigator, R.E. Knops, Principal Investigator, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NL64634_018_18
Record Dates: First submitted 2018-03-23; First posted 2018-04-12 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Ventricular Arrythmia
Keywords: subcutaneous implantable cardioverter defibrillator; Defibrillation testing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- S-ICD Implant with defibrillation test (No Intervention): Patients undergoing de novo S-ICD implantation including induction of VF and defibrillation testing post-implant
- S-ICD Implant without defibrillation test (Experimental): Patients undergoing de novo S-ICD implantation without induction of VF and defibrillation testing post-implant
  Interventions: Procedure: ommitence of defibrillation testing

INTERVENTIONS:
Procedure: ommitence of defibrillation testing — Induction of a ventricular arrhythmia to test proper arrhythmia detection and termination by the implanted device is omitted
  Arms: S-ICD Implant without defibrillation test

SUMMARY:
This study will test the hypothesis that implantation of a subcutaneous implantable cardioverter defibrillator (S-ICD) without performing a defibrillation test is non-inferior to S-ICD implant with a defibrillation test with regards to the primary endpoint failed first shock in a spontaneous arrhythmia episode when implant position is confirmed with PRAETORIAN score.

DETAILED DESCRIPTION:
Implantable Cardioverter Defibrillator (ICD) implant improves survival in patients with a higher risk for sudden cardiac death. There are 2 types of ICD available; transvenous ICD (TV-ICD) and subcutaneous ICD (S-ICD). During ICD implant, defibrillation testing (DFT) is performed to test functionality of the device. However, DFT can be associated with complications such as inability to convert, complications arising from general anaesthesia, prolonged resuscitation, stroke and death. Whereas DFT may be associated with complications, the benefit of DFT is debated as literature shows there is only a modest average effect of DFT, if any, on mortality, shock efficacy or safety. Recently it was shown in a randomized controlled trial called 'SIMPLE' that routine defibrillation testing of TV-ICDs at the time of implant does not improve shock efficacy or reduce arrhythmic death. For S-ICD there is only limited data available of the effect of DFT on S-ICD efficacy. Data have however shown that the conversion efficacy of the S-ICD is comparable to TV-ICD.

DFT is currently performed in standard S-ICD implants, but is omitted in specific cases. However, an alternative method to evaluate the correct position may be desired when omitting DFT. The PRAETORIAN Score is developed using computer modelling data on factors influencing defibrillation thresholds. The PRAETORIAN score represents the chance of a patient having an elevated defibrillation threshold and consequently failing a DFT or conversion of a spontaneous arrhythmia episode. The score was retrospectively validated in two studies with 180 and 321 patients.

It was reported that most S-ICD implants are performed under general anesthesia, however other anesthesia protocols are used as well. One of the most predominant factors to use general anesthesia is the performance of the DFT. If this is omitted, other anesthesia protocols may be a good option for many patients as well.

ELIGIBILITY:
Inclusion Criteria:

* Patients who meet current guidelines for ICD therapy and intent to undergo a de novo implant procedure for an S-ICD
* Patients must pass S-ICD screening per local routine
* Patients over 18 years of age, willing and capable to give informed consent
* Patients must be willing and capable of complying to follow up visits
* Patient must be eligible for either DFT strategy per physician discretion

Exclusion Criteria:

* Patient with a life expectancy shorter than 12 months due to any medical condition
* Patients known to be pregnant
* Patients with intracardiac thrombus
* Patients with atrial fibrillation without appropriate anticoagulation
* Patients likely to undergo heart transplant within 12 months
* Patients with LVAD
* Patients with other contra-indications for DFT per physician's discretion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 965 (Actual)
Dates: Start 2018-05-07 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Failed first appropriate shock in a spontaneous episode | 40 months
  Number of patients having experiences a failed first appropriate shock in a spontaneous arrhythmia episode

SECONDARY OUTCOMES:
DFT related complications | 24 hours or 30 days
  Number of patients experiencing DFT related complications occurring within 24h or 30 days after DFT
PRAETORIAN Score | up to 24 hours
  Implant position will be scored using the PRAETORIAN score
Pain post implant | 1-4 hours post implant
  Pain score measured with McGill questionnaire
Appropriate ICD therapy | 40 months
  Shocks given for VT or VF
Inappropriate ICD therapy | 40 months
  Shocks given for anything else than VT or VF
Overall DFT conversion success | 40 months
  The percentage of patients with at least one induced episode teminated by an S-ICD shock within five seconds post shock delivery
Successful DFT | 40 months
  A successful DFT is defined as conversion to SR or AF in less than 5 seconds from appropriate shock delivery.
Time to therapy | 40 months
  Time to therapy is the time between the start of VT or VF in a treated episode until the first shock in seconds.
Time to succesful therapy | 40 months
  Time to successful therapy is the time between the start of VT or VF until the first successful shock.
Shock efficacy | 40 months
  Percentage of appropriate shocks that was successfull
Conversion efficacy within 5 shocks in spontaneous episodes | 40 months
  Conversion efficacy within 5 shocks in spontaneous episodes
S-ICD related complications | 40 months
  S-ICD related complications requiring invasive intervention
MACE post DFT | 30 days
  Number of Major Adverse Cardiac Events after DFT procedure
Cardiac (pre-)syncope | 40 months
  Number of episodes of cardiac (pre-)syncope
Cardiac decompensation | 40 months
  Number of episodes of cardiac decompensation
Mortality | 40 months
  All cause mortality; arrhythmic death; cardiovascular death; unexplained death
Length of hospitalization | 40 months
  Length of hospitalization post implant (nights)
Device or lead repositioning | 40 months
  Number of procedures for device or lead repositioning
ICD related infection | 40 months
  Number of infections related to implanted ICD
Composite complications 30 days after implant | 30 days
  Number of patients experiencing complications occurring within 30 days after implant

CONTACTS AND LOCATIONS:
Overall Officials: Reinoud E Knops, MD, PhD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (32):
- United States (7):
  - Adventh Health System, Orlando, Florida
  - Emory University Hospital, Atlanta, Georgia
  - CorVita Science Foundation, Chicago, Illinois
  - Englewood Hospital and Medical Center, Englewood, New Jersey
  - Mount Sinai Beth Israel, New York, New York
  - Icahn School of Medicine at Mount Sinaï, New York, New York
  - Erlanger Health System, Chattanooga, Tennessee
- Germany (5):
  - Asklepios Kliniken, Hamburg
  - Universitätsklinikum Schleswig-Holstein, Kiel
  - Universitätsklinikum Schleswig-Holstein, Campus Lübeck, Lübeck
  - Universitätsklinikum Mannheim, Mannheim
  - Universitätsklinikum Würzburg, Würzburg
- Netherlands (11):
  - Flevoziekenhuis, Almere Stad
  - Academic Medical Center Amsterdam, Amsterdam
  - OLVG, Amsterdam
  - Albert Schweitzer Ziekenhuis, Dordrecht
  - Catharina Ziekenhuis, Eindhoven
  - UMCG, Groningen
  - Spaarne Gasthuis, Haarlem
  - Medisch Centrum Leeuwarden, Leeuwarden
  - St Antonius Ziekenhuis, Nieuwegein
  - Canisius Wilhelmina Ziekenhuis, Nijmegen
  - Isala Klinieken, Zwolle
- United Kingdom (9):
  - Basildon and Thurrock Univerity Hospital NHS Foundation Trust, Basildon
  - Blackpool Victoria Hospital NHS Foundation Trust, Blackpool
  - Royal Papworth Hospital NHS Foundation Trust, Cambridge
  - Heart and Chest Hospital NHS Foundation Trust, Liverpool
  - Barts Health NHS Trust of the Royal London Hospital, London
  - Manchester Heart Center, Manchester Royal Infirmary, Manchester
  - Oxford University Hospitals NHS Foundation Trust, Oxford
  - Sheffield Teaching Hospitals NHS Foundation Trust, Northern General Hospital, Sheffield
  - The Royal Wolverhampton NHS Trust, the New Cross Hospital, Wolverhampton

REFERENCES:
- [Background] Quast ABE, Baalman SWE, Betts TR, Boersma LVA, Bonnemeier H, Boveda S, Brouwer TF, Burke MC, Delnoy PPHM, El-Chami M, Kuschyk J, Lambiase P, Marquie C, Miller MA, Smeding L, Wilde AAM, Knops RE. Rationale and design of the PRAETORIAN-DFT trial: A prospective randomized CompArative trial of SubcutanEous ImplanTable CardiOverter-DefibrillatoR ImplANtation with and without DeFibrillation testing. Am Heart J. 2019 Aug;214:167-174. doi: 10.1016/j.ahj.2019.05.002. Epub 2019 May 16. PMID 31220775